CLINICAL TRIAL: NCT02434796
Title: A Mixed Methods Study to Test the Preliminary Effect of Together to End Violence Against Women (TEVAW): a Program to Address Intimate Partner Violence in Northern Tanzania
Brief Title: Study of the Preliminary Effect of TEVAW: a Program to Address Intimate Partner Violence in Northern Tanzania
Acronym: TEVAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: World Education, Inc. (Industry)
Responsible Party: Principal Investigator, Lisa J. Messersmith, Associate Professor, Boston University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SVRI49-WEI2014
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Gender-Based Violence; Gender; HIV
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Male Peer Groups (MPG) (Experimental): Women participate in savings groups and male partners participate in male peer group workshops on gender norms, IPV and HIV prevention. This intervention aims to improve knowledge and attitudes about the harms of IPV on women, men and children; the confidence to internalize positive masculine ideals (e.g. caring for one's family) and to challenge gender stereotypes (e.g. women are not equal to men); and the ability to formulate positive outcome expectations regarding IPV (intolerance of violence perpetrated by themselves or others) and healthy relationships with their spouses and communities.
  Interventions: Behavioral: Male Peer Groups
- Arm 2 MPG & Community Dialogues (Experimental): This arm will include women participants in savings groups, male peer groups and community dialogues. Village community leaders will engage in community dialogues on gender norms, IPV and HIV prevention.
  Interventions: Behavioral: Male Peer Groups and Community Dialogues

INTERVENTIONS:
Behavioral: Male Peer Groups — In Intervention Arm 1, male partners participate in male peer group workshops on gender norms, IPV and HIV prevention. Men's peer groups address gender inequality and transformation of gender power relations, positive masculinities and accountability of men in the perpetration of violence against women. This intervention aims to improve knowledge and attitudes among men about the harms of IPV on women, men and children; the confidence to internalize positive masculine ideals and to challenge gender stereotypes; and the ability to formulate positive outcome expectations regarding IPV and healthy relationships with their spouses and communities. Male peer group workshops will be conducted as a series of four workshops for a total of 24 hours spread out over a 5-month period.
  Arms: Arm 1 Male Peer Groups (MPG)
Behavioral: Male Peer Groups and Community Dialogues — Men participate in male peer group workshops as in Intervention Arm 1. In addition, village level community leaders engage in community mobilization/sensitization activities that include women members of savings groups and their male partners who participate male peer groups. Community dialogues focus on gender norms, IPV and HIV prevention. First, a one-day workshop for community leaders on topics similar to those raised in male peer group sessions. Second, trained community leaders facilitate community dialogues on IPV, HIV prevention, and gender norms with savings groups members and their male partners who participate in male peer groups. Each workshop will be a day-long event.
  Arms: Arm 2 MPG & Community Dialogues

SUMMARY:
Women in Tanzania suffer alarming rates of intimate partner violence (IPV) that has detrimental effects on mental and physical health including an increased risk of HIV infection. The investigators will use a cluster randomized control study design to conduct a preliminary evaluation study of TEVAW, an intervention that aims to improve gender equitable attitudes and to decrease tolerance of IPV among men and women in rural Tanzania. Nine villages will be randomly assigned into one of three study arms, each comprised of 150 partnered women and their co-resident male partners. Women in the comparison arm are currently exposed to World Education's savings and lending group intervention (known as LIMCA), in which they receive training on business skills, literacy, child nutrition and health, child protection, intimate partner violence (IPV) and HIV prevention. Women in Intervention Arm 1 will be exposed to LIMCA, while their male partners will participate in male peer group workshops that explore gender norms, IPV and HIV prevention issues. In Intervention Arm 2, men and women will receive the same treatment as Intervention Arm 1 and participate in community dialogues with community leaders to explore similar topics as the male peer groups. Our hypothesis is that study participants in Arm 2 will report improved gender equitable attitudes and lower intolerance of intimate partner violence than participants in Arm 1 and participants in the control group. Data will be collected at baseline and endline using a structured questionnaire with questions from three validated instruments that measure gender equitable attitudes and attitudes about IPV.

DETAILED DESCRIPTION:
Women in Tanzania suffer alarming rates of intimate partner violence (IPV) that has detrimental effects on mental and physical health including an increased risk of HIV infection. The investigators will use a cluster randomized control study design to conduct a preliminary evaluation study of TEVAW, an intervention that aims to improve gender equitable attitudes and to decrease tolerance of IPV among men and women in rural Tanzania. Nine villages will be randomly assigned into one of three study arms, each comprised of 150 partnered women and their co-resident male partners. A total of 450 women and their partners will be recruited for the study. Women in the comparison arm are currently exposed to World Education's savings and lending group intervention (known as LIMCA), in which they receive training on business skills, literacy, child nutrition and health, child protection, intimate partner violence (IPV) and HIV prevention. Women in Intervention Arm 1 will be exposed to LIMCA, while their male partners will participate in male peer group workshops that explore gender norms, IPV and HIV prevention issues. In Intervention Arm 2, men and women will receive the same treatment as Intervention Arm 1 and participate in community dialogues with community leaders to explore similar topics as the male peer groups. Our hypothesis is that study participants in Arm 2 will report improved gender equitable attitudes and lower intolerance of intimate partner violence than participants in Arm 1 and participants in the control group. Data will be collected at baseline and endline using a structured questionnaire with questions from three validated instruments that measure gender equitable attitudes and attitudes about IPV. The following are the specific aims of the study:

1. To test the feasibility, acceptability and proof of concept of two interventions (women's savings groups combined with male peer groups vs. women's savings groups combined with male peer groups and community dialogues) compared to a control group participating only in women's savings groups in Karatu District, Northern Tanzania.
2. To contribute to a better understanding of the attitudes, behaviors and social factors related to intimate partner violence through the exploration of cultural gender norms in Karatu District, Northern Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Married women, aged 18 and older, who live in Karatu District in Northern Tanzania with their male partners, who participate in the LIMCA program, are willing to participate, and provide informed consent.
* Male partners of women LIMCA members named above, aged 18 and older who live in Karatu District in Northern Tanzania, are willing to participate, and provide informed consent.

Exclusion Criteria:

* Women who are not partnered, who do not live in the study catchment area, who do not participate in the LIMCA program, and who do not provide informed consent
* Men who are not married or partnered, who do not live in the study catchment area; whose wives/partners do not participate in the LIMCA program, and who do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of men who report a husband is justified in beating his wife | 4 months
  For attitudes on IPV, men get the value of 1, if they agree that a husband is justified in hitting or beating his wife if she (a) burns the food; (b) argues with him; (c) goes out without telling him; (d) neglects the children; or (e) refuses to have sexual intercourse with him; men get a 0 if they do not agree with any of these statements.

SECONDARY OUTCOMES:
Difference in proportion of men who report gender-inequitable attitudes | 4 months
  We will measure men's gender-inequitable attitudes using an 18-item scale on attitudes toward gender norms in intimate relationships, known as the GEM (Gender Equitable Men). For each item listed on the GEM scale, men will report their level of agreement with Strongly Agree [=3], Agree [=2], Disagree [=1], and Strongly Disagree [=0]. Men will get a score ranging between 0 and 54, where 0 indicates that a man reports to maintain the most inequitable attitudes on gender and 54 indicates that he maintains the most equitable gender attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Messersmith, PhD, MPH, Principal Investigator — Boston University Center for Global Health and Development

REFERENCES:
- [Derived] Halim N, Steven Mzilangwe E, Reich N, Badi L, Simmons E, Servidone M, Bingham Holmes N 2nd, Kawemama P, Messersmith LJ. Together to end violence against women in Tanzania: Results of a pilot cluster randomized controlled trial to evaluate preliminary effectiveness of interpersonal and community level interventions to address intimate partner violence. Glob Public Health. 2019 Dec;14(12):1653-1668. doi: 10.1080/17441692.2019.1609062. Epub 2019 May 13. PMID 31084264